CLINICAL TRIAL: NCT05924880
Title: A Phase IIIb, Single Arm, Open-label, Multi-center Study on Durvalumab in Combination With Gemcitabine-based Chemotherapy as First Line Treatment for Chinese Patients With Unresectable Biliary Tract Cancers
Brief Title: A Phase 3b, Open-label, Multi-center Study on Durvalumab in Combination With Gemcitabine-based Chemotherapy as 1L Treatment for the Chinese Patients With Unresectable Biliary Tract Cancers (BTC)
Acronym: TopDouble
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D933AL00006
Record Dates: First submitted 2023-06-01; First posted 2023-06-29 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Biliary Tract Cancers
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- durvalumab in combination with gemcitabine-based chemotherapy (Experimental): single-arm
  Interventions: Drug: durvalumab

INTERVENTIONS:
Drug: durvalumab — Durvalumab 1500 mg as a 60-minute IV infusion in combination with gemcitabine-based chemotherapy Q3W. Upon completing chemotherapy, or discontinuing chemotherapy due to toxicity, durvalumab 1500 mg IV Q4W alone or in combination with gemcitabine.
  Other Names: IMFINZI

SUMMARY:
This is a Phase IIIb, open-label, single arm, multicentre study to assess the safety and efficacy of durvalumab in combination with investigator's choice of 3 different gemcitabine-based chemotherapy regimens in participants with aBTC with a WHO/ECOG PS of 0 to 2 at enrolment.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the safety of durvalumab combined with gemcitabine-based chemotherapy for participants with advanced BTC who have not previously received systemic therapy for advanced or metastatic BTC with WHO/ECOG PS of 0 to 2.

Eligible participants will received durvalumab in combination with gemcitabine-based chemotherapy(Gemcitabine+Oxalipatin; Gemcitabine+S1, Gemcitabine+Cisplatin) by investigator's choice.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 18 years at the time of screening.
2. Histologically confirmed, unresectable advanced or metastatic BTC including cholangiocarcinoma (intrahepatic or extrahepatic), gallbladder carcinoma.
3. Participants with previously untreated disease are eligible if presented with unresectable or metastatic BTC at initial diagnosis.
4. Prior curative intent treatment (surgery and, if given in the adjuvant setting, chemotherapy and/or radiation) is permitted, with recurrent disease >6 months. This includes participants with residual disease after surgery, who received chemotherapy, chemoembolization, or radiotherapy.
5. A WHO/ECOG PS of 0 to 2.
6. At least one lesion that qualifies as a RECIST 1.1 TL at baseline.
7. Participants with HBV infection (as characterised by positive HBsAg and/or anti-HBcAb with detectable HBV DNA, as per local laboratory standards) must be treated with antiviral therapy, as per institutional practice, to ensure adequate viral suppression (as per local laboratory standards) prior to enrolment. Participants must remain on antiviral therapy for the study duration and for 6 months after the last dose of study intervention. Participants who test positive for anti-HBc with undetectable HBV DNA (as per local laboratory standards) do not require antiviral therapy prior to enrolment. These participants will be tested at every cycle to monitor HBV DNA levels and initiate antiviral therapy if HBV DNA is detected (as per local laboratory standards). HBV DNA detectable participants must initiate and remain on antiviral therapy for the study duration and for 6 months after the last dose of study intervention.
8. Adequate organ and marrow function, as defined below.

   * Haemoglobin ≥ 9 g/dL
   * Absolute neutrophil count ≥ 1.5 × 109/L
   * Platelet count ≥ 100 × 109/L
   * Serum bilirubin ≤ 2.0 × ULN; this will not apply to participants with confirmed Gilbert's syndrome. Any clinically significant biliary obstruction should be resolved before enrolment.
   * ALT and AST ≤ 2.5 × ULN. For participants with hepatic metastases, ALT and AST ≤ 5 × ULN.
   * Calculated creatinine clearance > 50 mL/minute as determined by Cockcroft-Gault (using actual body weight) or 24-hour urine creatinine clearance. For chemotherapy regimens including carboplatin, oxaliplatin, or gemcitabine as monotherapy, the recommended threshold for calculated creatinine clearance is > 40 mL/minute as determined by Cockcroft-Gault (using actual body weight) or 24-hour urine creatinine clearance.
9. Must have a life expectancy of at least 12 weeks.
10. Body weight of > 30 kg.
11. Male or female.
12. Negative pregnancy test (serum) for women of childbearing potential.
13. Female participants must be one year post-menopausal (amenorrhoeic for 12 months without an alternative medical cause), surgically sterile, or using one highly effective form of birth control (a highly effective method of contraception is defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly). Women of childbearing potential must agree to use one highly effective method of birth control (see Appendix H for a complete list of highly effective birth control methods). They should have been stable on their chosen method of birth control from the time of screening throughout the total duration of the study and the drug washout period (90 days after the last dose of study intervention with durvalumab or 180 days after the last dose of durvalumab and gemcitabine-based therapy).

    - Non-sterilised male partners of a woman of childbearing potential must use a male condom plus spermicide (condom alone in countries where spermicides are not approved) throughout this period. Cessation of birth control after this point should be discussed with a responsible physician. Periodic abstinence, as well as the rhythm and withdrawal methods are not acceptable methods of birth control.
14. Male participants who intend to be sexually active with a female partner of childbearing potential must be surgically sterile or using an acceptable method of contraception (see Appendix H) from the time of screening throughout the total duration of the study and the drug washout period (90 days after the last dose of study intervention with durvalumab or 180 days after the last dose of durvalumab and gemcitabine-based therapy) to prevent pregnancy in a partner. Male participants must not donate or bank sperm during this same time period.

    - Female partners (of childbearing potential) of male participants must also use a highly effective method of contraception throughout this period.
15. Participant is capable of giving signed informed consent as described in Appendix A, Section A3 which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
16. Written informed consent from the participant has been obtained prior to any study-related procedures.

Exclusion Criteria:

1. Ampullary carcinoma.
2. As judged by the investigator, any evidence of diseases (such as severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diseases, active infection, active ILD/pneumonitis, serious chronic gastrointestinal conditions associated with diarrhoea, psychiatric illness/social situations), history of allogenic organ transplant, which, in the investigator's opinion, makes it undesirable for the participant to participate in the study or that would jeopardise compliance with the protocol.
3. Active or prior documented autoimmune or inflammatory disorders including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis], Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc). The following are exceptions to this criterion:

   * Participants with vitiligo or alopecia.
   * Participants with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement.
   * Any chronic skin condition that does not require systemic therapy.
   * Participants without an active disease in the last 5 years may be included but only after consultation with the study physician.
   * Participants with celiac disease controlled by diet alone.
   * Participants with ≥ Grade 2 lymphopenia will be evaluated on a case-by- case basis after consultation with the study physician
4. History of another primary malignancy, except for malignancy treated with curative intent and with no known active disease ≥ 5 years before the first dose of study intervention and of low potential risk for recurrence, basal cell carcinoma of the skin, squamous cell carcinoma of the skin or lentigo maligna that has undergone potentially curative therapy, or adequately treated carcinoma in situ without evidence of disease.
5. History of leptomeningeal carcinomatosis.
6. History of active primary immunodeficiency.
7. Known to have tested positive for HIV (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).
8. Participants co-infected with HBV (presence of HBsAg and/or anti-HBcAb with detectable HBV DNA, as per local laboratory standards) and HCV (presence of anti-HCV antibodies), or coinfected with HBV and HDV (presence of anti-HDV antibodies).
9. Persistent toxicities (CTCAE Grade > 2) caused by previous anticancer therapy; alopecia and vitiligo are excluded toxicities.

   * Participants with Grade ≥ 2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician.
   * Participants with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the study physician.
10. History of previous or current, brain metastases or spinal cord compression (including asymptomatic and adequately treated disease). Participants with suspected brain metastases at screening should have an MRI (preferred) or CT scan, each preferably with IV contrast of the brain prior to study entry.
11. Known allergy or hypersensitivity to any of the study intervention or any of the study intervention excipients.
12. Any concurrent chemotherapy, other than the one allowed in the study, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy) is acceptable.
13. Palliative radiotherapy with a limited field of radiation within 2 weeks of the first dose of study intervention, or radiotherapy with a wide field of radiation or radiotherapy affecting more than 30% of the bone marrow within 4 weeks before the first dose of study intervention. Prior locoregional therapy, such as radioembolization, is allowed as long as done more than 2 weeks prior.
14. Receipt of live attenuated vaccine within 30 days prior to the first dose of study intervention (see Appendix J). Enroled participants should not receive live vaccine while receiving study intervention and up to 30 days after the last dose of IP.
15. Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of IP. Minor surgery of isolated lesions for palliative intent is acceptable if performed more than 14 days prior to the first dose of IP.
16. Prior exposure to immune-mediated therapy including, but not limited to, other anti-CTLA-4, anti-PD-1, anti-PD-L1, and anti-PD-L2 antibodies, excluding therapeutic anticancer vaccines.
17. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, or topical steroids or local steroid injections (eg, intra-articular injection).
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
    * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
18. Receipt of the last dose of anticancer therapy (chemotherapy, targeted therapy, biologic therapy, or mAbs) within 28 days prior to the first dose of study intervention or 5 half-lives of the respective study intervention, whichever is longer.
19. Participation in another clinical study with a study intervention administered in the last 3 months.
20. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study, or during the follow-up period of an interventional study.
21. Prior randomisation or study intervention in a previous durvalumab clinical study, regardless of study intervention arm assignment.
22. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
23. Female participants who are pregnant or breastfeeding or male or female participants of reproductive potential who are not willing to use effective birth control from screening to 90 days after the last dose of study intervention with durvalumab or 180 days after the last dose of durvalumab and gemcitabine-based therapy.
24. Judgement by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
The incidence of Possible related adverse events(PRAE) Grade 3 or 4 | Within 6 months after the initiation of study intervention.
  The primary endpoint of this study is the incidence of Grade 3/4 PRAEs (CTCAE v5.0) of durvalumab combined with gemcitabine-based chemotherapy within 6 months of starting study intervention regardless of length of infusion. PRAEs are where the investigator answered yes to the question "Do you consider that there is a reasonable possibility that the event may have been caused by the investigational product?".

SECONDARY OUTCOMES:
Overall Survival(OS) | From first dose of study intervention until death, up to 67.9% OS maturity or at least 12 months after the last subject enrolled, which occurs first
  Overall Survival(OS) is defined as the time from the date of the first dose of study intervention until death due to any cause. The measures of interest are median Overall Survival(OS) and Overall Survival at 12 months(OS12).
Objective Response Rate (ORR) | From first dose of study intervention until disease progression or death (whichever occurs first), up to approximately 3 months after the last subject enrolled
  Objective Response Rate (ORR) is defined as the proportion of participants who achieved a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), assessed by BICR per RECIST Version 1.1.
Progression-free Survival (PFS) | From first dose of study intervention until disease progression or death (whichever occurs first), up to approximately 6 months after the last subject enrolled
  Progression-free Survival (PFS) is defined as the time from randomization to the first documented radiographic disease progression or death due to any cause, whichever occurs first, assessed by the Investigator per RECIST Version 1.1.
Disease Control Rate(DCR) | From first dose of study intervention until disease progression or death (whichever occurs first), up to approximately 6 months after the last subject enrolled
  Disease Control Rate(DCR) is defined as the percentage of participants who have a best objective response of confirmed CR or PR by Week 24/30 or who have demonstrated SD per RECIST 1.1 for at least 24/30 weeks following the start of treatment. The measure of interest is Disease Control Rate at 24 weeks(DCR24) and Disease Control Rate at 30 weeks(DCR30).
Duration of Response(DOR) | From first dose of study intervention until disease progression or death (whichever occurs first), up to approximately 6 months after the last subject enrolled
  Duration of Response(DOR) is defined as the time from the date of first documented response until the date of documented progression per RECIST 1.1 as assessed by the investigator or death due to any cause.
Duration of Treatment(DOT) | From first dose of study intervention until last dose or death (whichever occurs first), up to 67.9% OS maturity or at least 12 months after the last subject enrolled, which occurs first
  Duration of Treatment(DOT) is defined as time on study intervention.
Patient-reported Outcomes(PROs) | From first dose of study intervention until 90 days after last dose or death (whichever occurs first)
  Patient-reported outcome assessment is a general term referring to all outcomes and symptoms that are directly reported by the participant.
Incidence of treatment-emergent adverse events(AEs) | From first dose of study intervention until 90 days after last dose or death (whichever occurs first)
  Incidence of treatment-emergent adverse events(AEs), including possible related adverse events(PRAEs), adverse event of special interests(AESIs), immune-mediated adverse events(imAEs), and serious adverse events(SAEs).
Severity of treatment-emergent adverse events(AEs) | From first dose of study intervention until 90 days after last dose or death (whichever occurs first)
  Severity of treatment-emergent AEs, including possible related adverse events(PRAEs), adverse event of special interests(AESIs), immune-mediated adverse events(imAEs), and serious adverse events(SAEs).
Intervention/treatment of treatment-emergent adverse events(AEs) | From first dose of study intervention until 90 days after last dose or death (whichever occurs first)
  Intervention/treatment of treatment-emergent AEs, including possible related adverse events(PRAEs), adverse event of special interests(AESIs), immune-mediated adverse events(imAEs), and serious adverse events(SAEs).
Outcome of treatment-emergent adverse events(AEs) | From first dose of study intervention until 90 days after last dose or death (whichever occurs first)
  Outcome of treatment-emergent AEs, including possible related adverse events(PRAEs), adverse event of special interests(AESIs), immune-mediated adverse events(imAEs), and serious adverse events(SAEs).
Causality of treatment-emergent adverse events(AEs) | From first dose of study intervention until 90 days after last dose or death (whichever occurs first)
  Causality of treatment-emergent AEs, including possible related adverse events(PRAEs), adverse event of special interests(AESIs), immune-mediated adverse events(imAEs), and serious adverse events(SAEs).
Adverse Events(AEs) resulting in study intervention interruption and discontinuation | From first dose of study intervention until 90 days after last dose or death (whichever occurs first)
  Adverse Events(AEs) resulting in study intervention interruption and discontinuation

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Nanchang
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xiamen

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home